CLINICAL TRIAL: NCT06314256
Title: Clinical Evaluation of Hyaluronic Acid and Platelet Rich Fibrin Injection Efficacy in Interdental Papilla Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Baris Impram, Principal Investigator, Altinbas University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/218
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Interdental Papilla Loss
Keywords: interdental papilla loss; black triangle; interdental papilla reconstruction; hyaluronic acid; injectable platelet rich fibrin

STUDY DESIGN:
Intervention Model Description: A type of study used frequently in oral research: the mouth is divided into two or more subunits. Active and control (comparison) treatments are applied to the subunits (e.g., to the left and right sides).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be masked, which side of her/his mouth will be treated with either i-PRF or HA. The outcome assessor is blinded to the treatment modalities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable PRF (Active Comparator): i-PRF is produced by cenrifugation of patients own blood. Injection of 0.1-0.2 ml per interdental papilla 3 times with 3-week interval.
  Interventions: Biological: I-PRF Injection; Drug: Teosyal PureSense Global Action HA Injection
- Hyaluronic Acid (Active Comparator): Teosyal® Global Action PureSense. Composition: Cross-linked hyaluronic acid (HA): 25 mg/ml Lidocaine; 0,3%, (injection).
  Injection of 0.1-0.2 ml per interdental papilla 3 times with 3-week interval.
  Interventions: Biological: I-PRF Injection; Drug: Teosyal PureSense Global Action HA Injection

INTERVENTIONS:
Biological: I-PRF Injection — İnterdental papilla will be injected by i-PRF.
Drug: Teosyal PureSense Global Action HA Injection — Interdental papilla will be injected by Teosyal PureSense Global Action HA gel.

SUMMARY:
The goal of this clinical trial is to evaluate and compare the efficacy of injectable platelet rich fibrin (i-PRF) and hyaluronic acid (HA) in reconstruction of interdental papilla loss. The main questions it aims to answer are:

* How compareable are above mentioned two interventions (i-PRF&HA) in reconstruction of interdental papilla loss?
* Which treatment option is better accepted by patients? Which treatment option would patients be more satisfied with? Participants with multiple interdental papilla loss will be treated with both i-PRF and HA in split-mouth design. Researchers will compare two treatment options to see if black triangles caused by interdental papilla loss closes and if yes, for how long do they last.

DETAILED DESCRIPTION:
Nowadays, individuals give great importance to their appearance and dental aesthetics plays a key role in their personal appearance. Dental aesthetics is a combination of white and pink aesthetics formed by teeth and gums. The part of the gingival tissue that fills the triangular shaped spaces between the teeth is the interdental papilla. The presence of papillae in the teeth is closely related to the distance between the contact point between the teeth and the alveolar bone crest. Periodontal diseases, traumatic oral hygiene practices, incorrect orthodontic forces, incompatible restoration contour, the presence of diastema as a result of neighbouring teeth not being in contact, and tooth loss can cause loss of interdental papillae, resulting in the formation of gaps called black triangles. In addition to aesthetic problems, loss of interdental papillae can cause speech difficulties and food impaction.

Interdental papilla loss is one of the most important aesthetic periodontal difficulties and at the same time one of the most difficult problems to treat. Various surgical methods and flap designs have been proposed for the treatment and reconstruction of interdental papillae. However, current surgical methods have limited success and lack predictability, especially because the gingival papilla has a sensitive structure and less blood supply compared to other parts of the gingiva. Therefore, non-surgical methods have gained importance. As a result of the development of tissue engineering, dermal filling materials have started to be produced in recent years. Among these materials, hyaluronic acid (HA) is one of the basic components of connective tissue and especially its water binding/retention property makes it a determinant of tissue volume. HA enables the migration of fibroblast cells involved in collagen production and also acts as a liquid matrix where collagen and elastic fibres will proliferate. Due to these properties, Becker et al. first demonstrated in 2010 that it was possible to reconstruct a small area of interdental papilla loss in a minimally invasive and predictable manner using injectable HA gel. Subsequently, HA injections in interdental papil reconstructions have frequently been successfully reported in the literature.

Platelet Rich Fibrin (PRF) is an autologous, membrane-form product prepared by centrifugation of the patient's own blood. This fibrin matrix containing platelets, leukocytes and various growth factors is used especially in regenerative periodontal surgical operations. Injectable PRF (i-PRF), obtained by modifying the preparation protocol, forms a dynamic hydrogel by increasing the number of cells and releasing growth factors more frequently. I-PRF serves as a source of slow-release growth factors that help remodelling of the interdental papilla. Using data obtained through standardised photographs, the project will evaluate the effectiveness of area closure rates of black triangles caused by papilla loss over a 3-month period and measure patient feedback and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (without cardiovascular diseases, diabetes, thyroid diseases, auto-immune diseases)
* Patients with PPI 2 and PPI 3 papillae according to the Papillary Presence Index classification
* Probable pocket depth of 4 mm or less in the relevant area
* Plaque index and gingival index in the range of 0-1
* Neighbouring teeth in contact with each other in the relevant area
* Absence of any restoration in the relevant area
* Non-smoker
* No surgical periodontal treatment in the last 6 months
* For female subjects not pregnant or lactating
* No known allergy to hyaluronic acid

Exclusion Criteria:

* Not systemically healthy (with cardiovascular diseases, diabetes, thyroid diseases, auto-immune diseases)
* Diagnosed with periodontitis
* History of allergic reactions to hyaluronic acid
* Less than 2 mm keratinized tissue height in the relevant area
* Teeth crowding in relevant area
* Any kind of restoration (fillings, crowns, etc.) in the relevant area
* Smoker
* Ongoing orthodontic treatment
* Having parafunctional habits (bruxism, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Black Triangle Area | After the last injection: 1 month - 3 months
  Using standardized intraoral photographs, change in black triangle area in mm² will be measured
Intedental Papilla Reconstruction Rate | After the last injection: 1 month - 3 months
  Changes in Black Triangle Area given in percentage to the baseline values

SECONDARY OUTCOMES:
Patient Satisfaction Score | After the last injection: 3 months
  Patient satisfaction of each treatment option will be measured using Visual Analog Score (VAS).
Black Triangle Width | After the last injection: 1 month - 3 months
  Using standardized intraoral photographs, change in black triangle width in mm will be measured
Black Triangle Height | After the last injection: 1 month - 3 months
  Using standardized intraoral photographs, change in black triangle height in mm will be measured

OTHER OUTCOMES:
Correlation between Interdental Papilla Reconstruction Rate and Interdental Bone Crest-Interproximal Contact Point Distance | After the last Injection: 1 month-3 months
  Correlation between Interdental Papilla Reconstruction Rate(%) and Interdental Bone Crest-Interproximal Contact Point Distance(mm)
Correlation between Interdental Papilla Reconstruction Rate and Keratinised Tissue Thickness | After the last Injection: 1 month-3 months
  Correlation between Interdental Papilla Reconstruction Rate(%) and Keratinised Tissue Thickness(mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Altinbas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT06314256/Prot_SAP_000.pdf